CLINICAL TRIAL: NCT05827991
Title: A Randomized Controlled Trial of the Efficacy and Safety of 1565nm Non-ablative Fractional Laser on Treating Androgenic Alopecia
Brief Title: A Clinical Observation of 1565nm Non-ablative Fractional Laser in the Treatment of Androgenic Alopecia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: XijingH-PF-KY20222044-F-1
Record Dates: First submitted 2023-03-29; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-01

CONDITIONS: Androgenic Alopecia
Keywords: 1565nm Non-ablative Fractional Laser; Androgenic Alopecia; Treatment
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1565nm Non-ablative Fractional Laser (Experimental): 1565nm Non-ablative Fractional Laser
  Interventions: Device: 1565nm Non-ablative Fractional Laser
- Minoxidil (Active Comparator): Minoxidil for external use
  Interventions: Drug: 5% minoxidil external use
- 1565nm Non-ablative Fractional Laser combined with Minoxidil for external use (Active Comparator): 1565nm Non-ablative Fractional Laser combined with Minoxidil for external use
  Interventions: Device: 1565nm Non-ablative Fractional Laser combined with 5% minoxidil

INTERVENTIONS:
Device: 1565nm Non-ablative Fractional Laser — 1565nm Non-ablative Fractional Laser is used for treatment once every 2 weeks, a total of 10 times. 1565nm Non-ablative Fractional Laser uses square and rectangular light spots, and the size is adjusted according to the treatment area, which is about 8-16mm, 250-300spot, 10J/cm2.
  Arms: 1565nm Non-ablative Fractional Laser
Drug: 5% minoxidil external use — The method of use of 5% minoxidil tincture is for topical use on the scalp, 1 ml per time, 2 times per day.
  Arms: Minoxidil
Device: 1565nm Non-ablative Fractional Laser combined with 5% minoxidil — The two treatment mentioned above
  Arms: 1565nm Non-ablative Fractional Laser combined with Minoxidil for external use

SUMMARY:
1. Androgenic alopecia (AGA) is a clinically common non cicatricial, progressive hair follicle microminiaturization disorder that begins in puberty or after puberty. The latest epidemiological survey shows that the prevalence rate of males in China is about 21.3%. In 2021, Nature published an article stating that stress hormones can inhibit hair growth by regulating hair follicle stem cells. This research conclusion provides new evidence for the impact of stress on hair growth. The trend of receiving AGA patients in the investigators' outpatient department is increasing. How to provide rapid, safe, and effective treatment for AGA patients is currently a hot topic for clinicians.
2. Studies have shown that phototherapy can effectively improve androgenic alopecia, alopecia areata, and hair loss after chemotherapy, and promote hair growth. At the same time, phototherapy can also be adjusted by adjusting the expression of reductase genes and vascular endothelial growth factor genes, as well as some endogenous epidermal growth factors, such as fibroblast growth factor and insulin-like growth factor, are also upregulated, which can stimulate hair growth.

3.1565 nm non-ablative fractional laser has the effects of inhibiting sebaceous gland secretion of oil, regulating collagen metabolism, and delaying changes in scalp collagen after hair loss. Previous studies have confirmed that 1565 nm non-ablative fractional laser therapy for alopecia areata has a good effect. Its possible mechanisms include increasing local blood flow, stimulating growth factors and cytokines during hair growth. At the same time, in order to achieve low energy, safe, and effective treatment without the need for hair cutting, the investigators had for the first time improved the 1565 nm non non-ablative fractional laser treatment tool, removing the original sapphire crystal cooling contact. This improvement can make the treatment head fully fit the scalp, and the excitation beam acts vertically on the treatment area, reducing energy attenuation.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-40 years old, regardless of gender;
2. Clinical diagnosis of androgenic alopecia The diagnosis was based on the diagnostic criteria for androgenic alopecia in Clinical Dermatology, edited by Zhao Bian;
3. The patient agrees to participate in this trial and signs an informed consent form;
4. The scalp is free of bleeding, ulceration, infection, and other conditions that affect the visual field of laser surgery.

Exclusion Criteria:

1. Drugs that affect hair growth, including finasteride tablets, glucocorticoids, and vasoactive drugs, have been used within 6 months before treatment;
2. Those who undergo local scalp treatment within 3 months, including topical drugs, medical cosmetic treatment, etc;
3. Combined with severe damage to important organs such as heart, liver, kidney, and brain;
4. Symptomatic alopecia caused by other diseases, such as lupus erythematosus alopecia and folliculitis alopecia;
5. Scar constitution;
6. Patients with skin malignant tumors or precancerous lesions;
7. Pregnant or nursing;
8. Recent skin infections (such as viruses and bacteria);
9. Those who cannot persist in treatment and follow-up.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
hair mirror | 2 weeks
  Using a hair mirror, measure the hair density per unit area of the same part and field of view (the center of the longitudinal axis of the scalp and body), and calculate the number and density of hair per unit area.
BMI | 2 weeks
  weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Derpartment of Xijing Hospital, Xi'an, Shaanxi, China